CLINICAL TRIAL: NCT01955304
Title: A Single Center, Open-label, Randomized, Two-period Crossover Food Effect Study of Single Doses of Fruquintinib (HMPL-013) in Healthy Subjects
Brief Title: Food Effect Study of Single Dose of Fruquintinib (HMPL-013) in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012-013-00CH2
Record Dates: First submitted 2013-09-28; First posted 2013-10-07 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2013-05

CONDITIONS: Food Effect of Fruquintinib in Health Subjects
MeSH Terms: interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A-fasted dosing followed by fed dosing (Experimental): Experimental: Fasted dosing of fruquintinib followed by fed dosing; Dosing in the fasted state followed by fed dosing
  Interventions: Drug: fruquintinib
- B-fed dosing followed by fasted dosing (Experimental): Experimental: Fed dosing of fruquintinib followed by fasted dosing; Dosing in the fed state followed by fasted dosing
  Interventions: Drug: fruquintinib

INTERVENTIONS:
Drug: fruquintinib — Fruquintinib 4 mg capsule, 2 discrete single doses separated by 2-weeks
  Other Names: HMPL-013

SUMMARY:
This study will determine the effect of food on the pharmacokinetics (PK) of a single dose of 4mg fruquintinib in normal healthy subjects.

DETAILED DESCRIPTION:
This study will be an open-label, randomized, two-period, crossover PK food effect study of fruquintinib administered orally at 4mg. Subjects will be screened for eligibility up to 14 days prior to entry into the study.

For each of 2 study periods, subjects will be admitted to the clinical research unit (CRU) on the day before dosing and fast overnight (approximately 10 hours). On the morning of dosing for each of the 2 study periods, subjects will receive a single oral dose of 4 mg fruquintinib in either the fasted or fed state. Subjects will remain at the CRU for at least 120 hours after administration of study drug for collection of serial blood samples for pharmacokinetic (PK) analysis and safety monitoring. Subjects will return to the CRU for safety assessment for up to 336 hours postdose.

ELIGIBILITY:
Inclusion Criteria:

* Males , between 18 and 45 years of age, inclusive.
* Body mass index (BMI) within the range of 19 to 25 kg/m2, inclusive.
* In good health, determined by no clinically significant findings from medical history, physical examination, 12-lead ECG, and vital signs.
* Adequate hepatic, renal, heart, and hematologic functions
* Male subjects who are either sterile or agree to use, during the period from informed consent until 90 days following Study Completion, 1 of the following approved methods of contraception: a double barrier method (eg, male condom with spermicide, use by female sexual partner of an intrauterine device with spermicide, a female condom with spermicide, contraceptive sponge with spermicide, a diaphragm with spermicide, or use of a cervical cap with spermicide); a sterile sexual partner; a female sexual partner using an intravaginal system (eg,NuvaRing®); or a partner using an oral, implantable, transdermal, or injectable contraceptives.
* Able to comprehend and willing to sign an informed consent form (ICF).

Exclusion Criteria:

* Significant history or clinical manifestation of any significant metabolic/endocrine, allergic, dermatological, hepatic, renal, hematological, pulmonary, immune, cardiovascular, gastrointestinal, genitourinary, neurological, or psychiatric disorder(as determined by the Investigator).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator.
* History of stomach or intestinal surgery, nephrectomy, cholecystectomy or resection that would potentially alter absorption and/or excretion of orally administered drugs as determined by the investigator (appendectomy and/or hernia repair may be allowed).
* History or presence of an abnormal ECG, which, in the Investigator's opinion, is clinically significant.
* Diagnosis of alcoholism or drug addiction within 1 year prior to Period 1 Check-in.
* Participation in any other investigational drug study in which receipt of an investigational study drug occurred within 5 half-lives or 30 days, whichever is longer prior to informed consent.
* Use of any prescription medications or products within 14 days prior to Period 1 prior to informed consent.
* Use of any over-the-counter (OTC), non-prescription preparations (including vitamins, minerals, and phytotherapeutic, herbal, dietary supplements, or plant derived preparations) within 7 days prior to each study period Check-in.
* Use of alcohol-, grapefruit-, Seville orange-, or caffeine-containing foods, juices, or beverages within 72 hours prior to each study period Check-in.
* Use of known hepatic or renal clearance altering agents (eg, erythromycin, cimetidine, barbiturates, phenothiazines, or herbal/plant derived preparations such as St. John's Wort, etc.) for a period of 60 days prior to informed consent;
* Poor peripheral venous access.
* Donation of blood ≥ 250 mL from 30 days prior to informed consent until study completion, inclusive, or of plasma from 2 weeks prior to informed consent until study completion, inclusive.
* Receipt of blood products within 2 months prior to Period 1 Check-in;
* Blood pressure greater than 140/90 mmHg confirmed by repeat at Screening or at Period 1 Check-in.
* Any acute or chronic condition that, in the opinion of the Investigator, would limit the subject's ability to complete and/or participate in this clinical study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
• To determine the effect of food on the PK of a single dose of 4mg fruquintinib in normal healthy subjects. | Planned Enrollment/Screening Duration: Approximately 2 weeks. Length of Each Confinement: Approximately 7days prior to dose until approximately 120 hours postdose. Planned Study Conduct Duration: Approximately 6 weeks
  Blood samples for PK analysis of serum fruquintinib levels will be collected for a 2-week period following each of 2 doses.

SECONDARY OUTCOMES:
• To assess the safety and tolerability of single doses of 4mg fruquintinib | Planned Enrollment/Screening Duration: Approximately 2 weeks. Length of Each Confinement: Approximately 7days prior to dose until approximately 120 hours postdose. Planned Study Conduct Duration: Approximately 6 weeks
  Safety will be assessed by physical exam, clinical laboratory evaluations and ECGs.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Qian H, Fan S, Li K, Sai Y, Su W, Chen Q, Liu Y, Li T, Wang W, Jia J, Yu C, Liu Y. Effects of a High-fat Meal on the Pharmacokinetics of the VEGFR Inhibitor Fruquintinib: A Randomized Phase I Study in Healthy Subjects. Clin Ther. 2019 Aug;41(8):1537-1544. doi: 10.1016/j.clinthera.2019.05.014. Epub 2019 Jul 1. PMID 31272709